CLINICAL TRIAL: NCT01818700
Title: A Multicenter, Phase IV, Interventional Study to Assess the Efficacy and Safety of NORSPAN® (Buprenorphine) in Korean Patients With Spinal Disorders (NOBLE)
Brief Title: An Interventional Study to Assess the Efficacy and Safety of Buprenorphine in Korean Patients With Spinal Disorders
Acronym: NOBLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BUP12-KR-401
Record Dates: First submitted 2012-10-18; First posted 2013-03-26 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Disorder
MeSH Terms: conditions — Spinal Diseases | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm-Norspan patch (Buprenorphine) (Other): This trial is single arm with Norspan patch. Treatment with NORSPAN Ò will be started from 5 μg/h (1 patch a week) for 2 weeks, and proper titration (up-titration) will be allowed at visit 2(wk 2) and at visit 3(wk 4) according to the investigator's decision. The up-titration will be considered by investigator's judgement as follows; (1) if the rescue medication was used more than 2 times per day, on average or (2) based on the daily average NRS(Numeric Rating Scale), if the NRS was changed to worsen since the previous visit, (3) Investigator's judgement by considering any titration needed situation (e.g. dose, frequency of rescue medication).
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — 8weeks treatment with Norspan®(Buprenorphine)

SUMMARY:
The purpose of this study is to assess the pain reduction rate after 8 weeks treatment of NORSPAN® from baseline.

And secondary purpose are: pain reduction rate after 4 weeks treatment from baseline(week 0) the EQ-5D, the pain and sleep questionnaire, physician's overall satisfaction subject's overall satisfaction, and safety

DETAILED DESCRIPTION:
Upon providing written informed consent, subject will be screened in the study and assessment will be performed at that time such as safety laboratory assessments, physical examination, vital sign, medical history taking, 24 hours pain intensity score, EQ-5D, pain and sleep questionnaire, physician's overall satisfaction and subject's overall satisfaction.

If patient is eligible in inclusion/exclusion criteria at the time of visit 1, the patient will receive treatment with NORSPAN®.

Treatment with NORSPAN® will be started from 5 μg/h (1 patch a week) for 2 weeks, and proper titration (up-titration) will be allowed at visit 2(wk 2) and at visit 3(wk 4) according to the investigator's decision.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old or above male or female Korean patients
* Patients who have spinal disorders related pain
* Patients who had been treated with weak opioids and/or NSAIDs before study participation
* Patients who have moderate to severe pain intensity
* Naïve patients for Buprenorphine (Naïve patient are defined as those who had not been treated with Buprenorphine for 90 days)
* Patients who signed a written informed consent form

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. UNLESS they are:

  * women whose partners have been sterilized by vasectomy or other means
  * using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
* Patients with known hypersensitivity to buprenorphine or to any of the excipients
* Patients with severely impaired respiratory function or respiratory depression status
* Patients concurrently receiving MAOIs or who have received MAOIs within the previous two weeks
* Patients with convulsive disorders, head injury, shock, a reduced level of consciousness of uncertain origin, intracranial lesions or increased intracranial pressure, or in patients with severe hepatic impairment
* Patients with biliary tract disorders
* Patients known to have, or suspected of having a history of drug abuse
* Patients with history of opioid or drug dependence
* Patients who are concurrently taking other CNS depressants or muscle relaxants that may cause respiratory depression, hypotension, profound sedation or potentially result in coma.
* Patients who are taking Buprenorphine or strong opioid.
* Any situation where Buprenorphine is contraindicated
* Major surgery within 1 month prior to screening or planned surgery Mainly pain originated other than spinal disorders disease
* Non-malignant patients or cancer patients who are receiving any oncology treatment that could affect the measure of pain control
* With a disability that may prevent the patient from completing all study requirements and in particular, interfere with 24hrs pain intensity score
* Clinically significant impairment of cardiovascular, respiratory and renal function
* Patient who needs acute dose titration or whose pain intensity fluctuate significantly in a short period according to investigator's judgment
* Having used other investigational drugs at the time of enrollment, or within 30 days of enrollment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Whan Eoh, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Duration of study: from 16 Oct. 2012 to 28 Jun 2013
Pre-assignment Details: This study is single arm for Norspan(buprenorphine) patch. Treatment with NORSPAN will be started from 5 μg/h for 2 weeks, and proper titration(up-titration) will be allowed at visit 2(wk 2) and at visit 3(wk 4) according to the investigator's decision. judgement by considering any titration needed situation.
Groups:
- Single Arm - Norspan Patch (Buprenorphine): This study is single arm for Norspan(buprenorphine) patch. Treatment with NORSPAN Ò will be started from 5 μg/h (1 patch a week) for 2 weeks, and proper titration (up-titration) will be allowed at visit 2(wk 2) and at visit 3(wk 4) according to the investigator's decision. The up-titration will be considered by investigator's judgement as follows; (1) if the rescue medication was used more than 2 times per day, on average or (2) based on the daily average NRS(Numeric Rating Scale), if the NRS was changed to worsen since the previous visit, (3) Investigator's judgement by considering any titration needed situation (e.g. dose, frequency of rescue medication).
Period: Overall Study
Arm/Group | Single Arm - Norspan Patch (Buprenorphine)
Started | 245 (The No. of enrolled patients)
Safety Set | 241 (4 subjects were not study drug administered.)
FAS Set | 210 (31 subjects excluded from FAS due to no assessment of primary efficacy(26) and IC/EC violation(5).)
PP Set | 105 (105 subjects excluded from PP set due to various reasons.)
Completed | 141 (104 subjects dropped out this study prior to study completion.)
Not Completed | 104
Not completed — Adverse Event | 67
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 27
Not completed — Protocol Violation | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The No. of enrolled patients: 245 No. of patient for Safety set: 241(excluded 4 patients who were not applied study drug) No. of patient for FAS analysis set: 210 No. of patient for PP analysis set: 105
Groups:
- Norspan Patch (Buprenorphine): Trade name is Norspan. Buprenorphine 5μg/h, 10 μg/h, 20 μg/h patches will be used (4 patches a box). Patch will be administered every 7th day.
  Buprenorphine: 8weeks treatment with Norspan®(Buprenorphine)
Arm/Group | Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 241
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 63.51 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167
  Male | 74
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 241

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Intensity* at Week 8 of Treatment With the Study Drug From Baseline
Description: NRS-Pain scale assessed the severity of a subject's lower back pain on a scale of 0 (No pain) and 10 (Worst possible pain). NRS-Pain scale: Change = mean score at Week 8/ET minus mean score at Baseline.
Time Frame: 8 weeks
Population: FAS set: 210. Missing values were imputed by LOCF FAS included the data obtained from all subjects who had at least one dose of the study drug and had data of at least one primary efficacy endpoint assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Single Arm-Norspan Patch (Buprenorphine): This study is single study with buprenorphine. Treatment with NORSPAN Ò will be started from 5 μg/h (1 patch a week) for 2 weeks, and proper titration (up-titration) will be allowed at visit 2(wk 2) and at visit 3(wk 4) according to the investigator's decision. The up-titration will be considered by investigator's judgement as follows; (1) if the rescue medication was used more than 2 times per day, on average or (2) based on the daily average NRS(Numeric Rating Scale), if the NRS was changed to worsen since the previous visit, (3) Investigator's judgement by considering any titration needed situation (e.g. dose, frequency of rescue medication).
Arm/Group | Single Arm-Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 210
units on a scale | -1.65 (1.96)
Statistical Analysis 1: Comparison: Single Arm-Norspan Patch (Buprenorphine); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; The primary endpoint will be the actual reduction rate of pain intensity (0 -10) score at 8 weeks. It will be analyzed by using paired t-test; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-10 to 10], Standard Deviation 1.96

2. Secondary Outcome: Change of Pain Intensity at 4 Week of Treatment With Study Srug From Baseline.
Description: NRS-Pain scale assessed the severity of a subject's lower back pain on a scale of 0 (No pain) and 10 (Worst possible pain). NRS-Pain scale: Change = mean score at Week 4/ET minus mean score at Baseline.
Time Frame: 4 weeks
Population: FAS set: 210. Missing values were imputed LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm-Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 210
units on a scale | -1.26 (1.71)

3. Secondary Outcome: Change in Quality of Life at 8 Week of Treatment With Study Drug From Baseline
Description: The Euroqol Health Survey (EQ-5D, 3-level) was completed on five dimensions (mobility, self care, usual activities, pain/discomfort and anxiety/depression) to measure health-related quality of life on a scale from 0-1. A higher score indicates better quality of life.
  EQ-5D score = 1 - 0.081 - (relevant score by level for the relevant item)-0.269 (only if there is at least one level 3).
  Table of scores by level for EQ-5D items mobility(level 1=0, level2=0.069,level 3=0.314), self care(level 1=0, level2=0.104,level 3=0.214), usual activities(level 1=0, level2=0.036,level 3=0.094), pain/discomfort (level 1=0, level2=0.,level 3=0.386) and anxiety/depression(level 1=0, level2=0.071,level 3=0.236).
Time Frame: 8 weeks
Population: FAS set: 210. Missing values were imputed by LOCF. Even though 210 subjects at Visit 1, baseline were assessed EQ-5D questionnaire, At visit 4(8weeks), 153 subjects were assessed EQ-5D questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm - Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 153
units on a scale | 0.18 (0.31)

4. Secondary Outcome: Change of EQ-VAS at 8 Weeks of Treatment With Study Drug From Baseline.
Description: EQ-5D Visual Analogue Scale (VAS) in rates the participant's overall health status using values from 0 (worst imaginable) to 100 (best imaginable).
Time Frame: 8 week
Population: FAS set: 210. Missing values were imputed by LOCF. Even though 210 subjects were assessed EQ-VAS at visit 1(baseline), 153 Subjects were assessed EQ-VAS at visit 4(8week)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm - Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 153
units on a scale | 10.55 (24.76)

5. Secondary Outcome: Clinician Global Impression of Change(CGIC)
Description: Number of clinician with categorical change in overall status. CGIC: a clinician-rated instrument assessing change in clinician's overall status from baseline, on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: 8weeks
Population: FAS set: 210. Missing values were imputed by LOCF.
Measure: Number; unit: participants
Arm/Group | Single Arm - Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 210
participants
  Very much improved | 16
  Much improved | 63
  Minimally improved | 55
  No change | 68
  Minimally worse | 8
  Much worse | 0
  Very much worse | 0

6. Secondary Outcome: Patients Global Impression og Change(PGIC)
Description: Number of clinician with categorical change in overall status. PGIC: a participant-rated instrument assessing change in patient's overall status from baseline, on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: 8 week
Population: FAS set: 210. Missing values were imputed by LOCF.
Measure: Number; unit: participants
Arm/Group | Single Arm - Norspan Patch (Buprenorphine)
Number analyzed (Participants) | 210
participants
  Very much improved | 12
  Much improved | 60
  Minimally improved | 57
  No change | 71
  Minimally worse | 10
  Much worse | 0
  Very much worse | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Norspan Patch (Buprenorphine)
Serious Adverse Events (participants affected / at risk) | 1/241
Other Adverse Events (participants affected / at risk) | 143/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norspan Patch (Buprenorphine) (N=241)
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — This event was not an ADR. The relevant subject underwent a surgery due to this AE and the final outcome was recovered.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norspan Patch (Buprenorphine) (N=241)
Nausea (Gastrointestinal disorders) | 71 (77)
Vomiting (Gastrointestinal disorders) | 35 (36)
Constipation (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 50 (52)
Headache (Nervous system disorders) | 14 (14)
Somnolence (Nervous system disorders) | 6 (7)
Lethargy (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (24)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Chest discomfort (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Sleep disorder (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Polydipsia (Metabolism and nutrition disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Lacrimal disorder (Eye disorders) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No